CLINICAL TRIAL: NCT01384773
Title: Increasing CrossLinking of Corneal Collagen in Eyes With Progressive Keratoconus or Ectasia
Brief Title: Progressive Keratoconus or Ectasia Treatment Plan
Status: No longer available | Type: Expanded Access
Sponsor: Stephen Trokel (Other)
Responsible Party: Sponsor-Investigator, Stephen Trokel, Professor of Clinical Ophthalmology, Columbia University
Organization: Columbia University (Other)
Other Study IDs: AAAF0594
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus; Ectasia
Keywords: Keratoconus; Ectasia; UVA light; riboflavin; post-LASIK (laser in situ keratomileusis); pellucid marginal degeneration; irregular astigmatism
MeSH Terms: conditions — Keratoconus; Dilatation, Pathologic | interventions — Ophthalmic Solutions

INTERVENTIONS:
Other: Riboflavin Solution — This solution is used to saturate the corneal stroma prior to its photochemical activation by the IROC UV-X illuminator.
  Other Names: Medio-Cross Riboflavin 0.1% ophthalmic solution
Device: UV-X Illumination System — IROC UV-X irradiation system creates a uniform 11 mm circle of UVA light that is focused onto the corneal surface. This system is designed to irradiate the riboflavin saturated cornea with a uniform field of UVA light centered at 365 nm.
  Other Names: IROC UV-X System

SUMMARY:
Keratoconus and pellucid marginal degenerations are genetically based ocular conditions and post surgical ectasia is an iatrogenic condition. These diseases are characterized by weakening of the front part of the eye that causes thinning and distortion. This distortion results in unevenness of the cornea and produces progressive near-sightedness and irregularity, which causes loss of vision when using eyeglasses. When eyeglasses fail to give enough vision, the the investigators use rigid contact lenses to create an artificial front eye surface. This improves visual acuity in many patients although they eventually fail either because they cannot be tolerated or the surface irregularity has become so severe that they are rejected. At this stage there is usually thinning and loss of clarity of the eye.

There has been no treatment for this other than corneal transplantation, a complex surgical procedure with a significant complication rate and a delay in visual recovery. The treatment the investigators wish to perform strengthens the front of the eye by a chemical reaction using light and riboflavin. This technique has been studied over a decade and is widely used throughout the world. The FDA approved multicenter American clinical study is being analyzed in anticipation of its submission to the FDA for PreMarket approval. Because this is a progressive condition, the investigators wish to be able to offer this on a limited basis to patients in need with vision loss.

Any treatment that can delay or prevent corneal transplantation is of great benefit. The investigators believe the evidence is compelling that this treatment is the sole alternative to surgical transplantation.

DETAILED DESCRIPTION:
Potential candidates will undergo a complete eye examination to determine their eligibility for treatment. Eligible subjects will be prepared for treatment in accordance with the instructions for use in the UV-X™ Illumination System Operator's Manual, including the administration of the riboflavin and preoperative medications (e.g. topical anesthetics). Prescriptions for postoperative medications and written postoperative instructions will be given to each subject and reviewed prior to discharge. All subjects will have follow-up examination at 1 day, 1 week, 3 month and 6 month.

ELIGIBILITY:
Inclusion Criteria:

Subjects who have one or both eyes that meet all of the following criteria will be considered candidates for this treatment:

For Keratoconus and Post Refractive Surgery Ectasia:

1. 16 years of age or older
2. Having a diagnosis of keratoconus with one or more of the following changes over a period of 24 months or less.

   1. An increase of > 1.00 D in the steepest keratometry value (or sim K)
   2. An increase of > 1.00 D in regular astigmatism evaluated by subjective manifest refraction
   3. A myopic shift (decrease in the spherical equivalent) of > 0.50 D on subjective manifest refraction
   4. Documented decrease in visual acuity associated with irregular astigmatism and topographic features of ectasia.
3. Presence of central or inferior steepening on the Pentacam map.
4. Axial topography consistent with keratoconus
5. Slit lamp findings associated with keratoconus must be documented:

   * Fleischer ring
   * Vogt striae
   * Corneal thinning
   * Corneal scarring
6. Contact Lens Wearers Only: Removal of contact lenses are required prior to the screening
7. Signed written informed consent

Exclusion Criteria:

All subjects meeting any of the following criteria will be excluded from this treatment:

1. No evidence of progression.
2. Excessively thin corneas.
3. Previous ocular condition in the eyes to be treated that may predispose the eye for future complications, for example:

   1. History of corneal disease (e.g., herpes simplex, herpes zoster keratitis, recurrent erosion syndrome, corneal melt, corneal dystrophy, etc.)
   2. Clinically significant corneal scarring in the proposed treatment zone
4. A history of chemical injury or delayed epithelial healing in the eye(s) to be treated.
5. A known sensitivity to treatment medications
6. Patients with a current condition that, in the treating physician's opinion, would interfere with or prolong epithelial healing.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Trokel, MD, Principal Investigator — Columbia University, Department of Ophthalmology, College of Physicians and Surgeons
Locations (1):
- Edward Harkness Eye Institute-Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Wittig-Silva C, Whiting M, Lamoureux E, Lindsay RG, Sullivan LJ, Snibson GR. A randomized controlled trial of corneal collagen cross-linking in progressive keratoconus: preliminary results. J Refract Surg. 2008 Sep;24(7):S720-5. doi: 10.3928/1081597X-20080901-15. PMID 18811118